CLINICAL TRIAL: NCT06942793
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Active-Controlled Study to Evaluate the Efficacy and Safety of Treatment With CsA-PG Ophthalmic Gel in Dry Eye Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of Treatment With CsA-PG Ophthalmic Gel in Dry Eye Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKY-CSA-202401
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1 drop each time, bilaterally once daily
  Interventions: Drug: CsA-PG Ophthalmic Gel
- Control group (Placebo Comparator): 1 drop each time, bilaterally once daily
  Interventions: Drug: CsA Ophthalmic Gel

INTERVENTIONS:
Drug: CsA-PG Ophthalmic Gel — Administer to eyes
  Arms: Experimental group
Drug: CsA Ophthalmic Gel — Administer to eyes
  Arms: Control group

SUMMARY:
This is a phase III, multicenter, randomized, double-masked, Active-controlled design. The aims to confirm previous findings of the efficacy and safety of CsA-PG Ophthalmic Gel by comparing it to CsA Ophthalmic Gel for treating dry eye symptoms.

DETAILED DESCRIPTION:
396 subjects will be enrolled (198 in each treatment group). Subject selection will be conducted during a 14-day run-in period before randomization. After the screening, subjects will receive lubricant eye drops (Refresh Tears®, Carboxymethylcellulose Sodium (0.5%)) treatment bilaterally BID for 14 days. Eligible subjects will be randomized (1:1) and receive the experimental drug or control drug , administered bilaterally once daily for 84 days.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age, male or female;
2. Provide written informed consent;
3. Have a reported history of dry eye for at least 6 months before Visit 1;
4. Have a clinical diagnosis of bilateral dry eye disease, including all of the following scored in at least one eye at both Visits 1 and 2;

   1. Corneal fluorescein staining score in either inferior, superior, or central zone ≥ 2
   2. Schirmer Tear Test score (STT, anesthetized) of ≤ 10 mm and ≥ 1 mm
   3. Have an Eye Dryness Score (EDS; Visual Analogue scale, VAS) ≤80 and ≥40

Exclusion Criteria:

1. Clinical diagnosis or history of any clinically significant ocular diseases/disorders (e.g., age-related maculopathy that requires treatment and/or in the opinion of the Investigator may interfere with study parameters in Visit 1 and/or Visit 2;
2. Any active ocular or systemic infection (e.g., bacterial, viral, or fungal) at Visit 1 and/or Visit 2;
3. Any active ocular inflammation (e.g., iritis, uveitis, allergic conjunctivitis) at Visit 1 and/or Visit 2;
4. Any conjunctival scarring history (Such as with irradiation, alkali burns, Steven Johnson syndrome, Sjogren's syndrome, cicatricial pemphigoid) or destruction of conjunctival goblet cells (e.g., neurotrophic keratitis, vitamin A deficiency) before Visit 1;
5. Have worn contact lenses within 14 days of Visit 1 or anticipate using contact lenses during the study;
6. Have any refractive surgery and/or any other ocular surgical procedure within 3 months before Visit 1; or have any ocular surgical procedure scheduled to be conducted during the study period;
7. Have eyelid surgery within 6 months before Visit 1 or planned eyelid surgery during the study period;
8. Have Nd:YAG (neodymium-doped yttrium aluminum garnet) laser capsulotomy within 6 months before Visit 1;
9. Have used temporary (i.e., collagen) punctual plugs within 3 months before Visit 1 or anticipate their use during the study period;
10. Have permanent punctual plugs inserted or have surgical punctual occlusion before Visit 1 or anticipate any such event during the study period;
11. Use any of the following treatments in the period indicated before Visit 1 or anticipate their use at any time during the study.

    Topical medications（30 days prior to Visit 1）:
    * Restasis®, Cequa™, Tyrvaya, Eysuvis, Xiidra
    * Topical ophthalmic non-steroidal anti-inflammatories
    * Topical ophthalmic corticosteroids
    * Topical ophthalmic autologous serum Exceptions: demulcent ophthalmic drops (e.g., OCCT artificial tears) may be used until Screen Visit 1, but these must be discontinued after screening.

    Systemic medication (30 days before Visit 1):

    Any systemic medication known to cause ocular drying (e.g., antidepressants, beta blockers) except if it was taken on a stable dosing regimen for at least 30 days before Visit 1 and is expected to be taken on the same regimen throughout the study period. The known systemic medications that can cause ocular drying include:
    * antihistamines, antidepressants, bronchodilators, antiarrhythmics
    * anti-Parkinson's disease drugs, antipsychotics, antitussives, anticongestants
    * adrenoceptor blockers, thiazide diuretics, anti-leprosy drugs, antimalarials, antineoplastics anxiolytics/sleeping agents, herbs and vitamins, calcium modulators
    * Corticosteroids (e.g., systemic steroids including intravenous, intramuscular, intraarticular, and oral steroids; facial topical steroids; dermatological steroids with high potency or large treatment areas)
    * Cyclosporine and any other immunosuppressor
    * Other medications that can impact dry eye disease favorably or not include various analgesics, including opiates, cannabinoids, omega-3 dietary supplements, and other agents. Such meds should be continued on study only if that represents a continuation of an unavoidable and unchanged regimen of treatment for a disease that is not otherwise excluded

    Non-medicine treatment (30 days before Visit 1):
    * LipiFlow® or other similar meibomian gland dysfunction (MGD) therapy;
    * Eye mask with heat or steam and any other warming method of the eyelid (e.g., warm towel application);
    * Intense pulsed light treatment;
    * Bandage contact lenses or scleral contact lenses;
    * Route eyelid cleaning;
    * Any other treatment that will relieve dry eye symptoms and signs.
12. Have a severe/serious systemic disease, chronic illness, or uncontrolled medical condition including, but not limited to, severe cardiopulmonary disease, poorly controlled hypertension, poorly controlled diabetes, and/or clinically significant (CS) hematologic, renal, or liver disease that in the opinion of the Investigator could interfere with study assessments or limit compliance;
13. Be a woman who is pregnant, nursing, or planning a pregnancy;
14. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 5 (or early termination visit) if of childbearing potential. The non-childbearing potential is defined as a woman who is permanently sterilized (e.g., has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is post-menopausal (i.e., without menses for 12 consecutive months);
15. Be a woman of childbearing potential who is not using an acceptable means of birth control during the study period and 30 days after the end of the study. Acceptable methods of contraception include hormonal (e.g., oral, implantable, injectable, or transdermal contraceptives), mechanical (e.g., spermicide in conjunction with a barrier such as a diaphragm or a condom), intrauterine device (IUD), or surgical sterilization of partner. For non-sexually active females, abstinence might be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use acceptable birth control as defined above for the remainder of the study;
16. Have a known hypersensitivity or contraindication to the investigational products (IPs) or their components;
17. Have a condition or be in a situation that the Investigator felt may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study (e.g., any planned procedure or surgery during the study period);
18. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days before Visit 1;
19. In the opinion of the Investigator, be unable or unwilling to comply with the study protocol, including participation in all study assessments, visits, and dosing, or be unable to instill eye drops successfully.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Eye Dryness Score(EDS) | 84 days
  The mean change from baseline in EDS (Eye Dryness Score) at the 84 days , with EDS assessment performed using a Visual Analogue Scale (VAS). The VAS score employs a 0 to 100-point scale (0 = no symptoms; 100 = extreme severity/intolerable discomfort), where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Total Corneal Staining Score(TCSS) | 84 days
  The proportion of patients achieving complete resolution of total corneal staining (TCSS= 0 ) at Day 84.TCSS is scored on a 0-to-20-point scale, higher numerical values correlate with increased severity of corneal damage.
Schirmer Tear Test (STT) | 84 days
  At day 84, the proportion of patients improved by ≥ 10 mm from baseline.

IPD SHARING:
Plan to Share IPD: Undecided